CLINICAL TRIAL: NCT05317741
Title: A Phase 1, First-in-human, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Food Effect, and Pharmacodynamics Following a Single Oral Dose of IA-14069 in Healthy Male Subjects
Brief Title: SAD Study of IA-14069
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ILAb Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: IA-14069_1a
Record Dates: First submitted 2021-10-27; First posted 2022-04-08 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- A mg IA-14069 or Placebo (Experimental)
  Interventions: Drug: IA-14069; Drug: Placebo
- B mg IA-14069 or Placebo (Experimental)
  Interventions: Drug: IA-14069; Drug: Placebo
- C mg IA-14069 or Placebo (Experimental): Period 1: Fasted condition → Period 2: Fed condition
  Interventions: Drug: IA-14069; Drug: Placebo
- D mg IA-14069 or Placebo (Experimental)
  Interventions: Drug: IA-14069; Drug: Placebo
- E mg IA-14069 or Placebo (Experimental)
  Interventions: Drug: IA-14069; Drug: Placebo

INTERVENTIONS:
Drug: IA-14069 — Subjects received IA-14069 tablet orally on Day 1.
Drug: Placebo — Subjects received matching placebo tablet orally on Day 1.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, food effect, and pharmacodynamics following a single oral dose of IA-14069 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the ICF.
2. Male subjects, ≥ 18 to ≤ 55 years of age at the time of signing the ICF.
3. Overtly healthy as determined by medical evaluation including medical history, physical examination and clinical laboratory tests.
4. Body mass index (BMI) within ≥ 18.0 to ≤ 32.0 kg/m2 and body weight not less than 50 kg.
5. Pulse rate between 40 and 100 beats per minutes (bpm)
6. A 12-lead ECG consistent with normal cardiac conduction and function, including:

   * Sinus rhythm
   * QTc interval of ≤ 450 milliseconds (QT interval corrected using Fridericia correction method [QTcF])
   * QRS interval of ≤ 120 milliseconds
   * PR interval ≤ 220 milliseconds
   * Morphology consistent with healthy cardiac conduction and function
7. Non-smoker or ex-smoker for > 6 months.
8. Agree to use contraception (Appendix 1) during the treatment period and for at least 90 days after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

1. Resting BP systolic or diastolic > 140/90 mmHg or < 90/45 mmHg. Subjects BP may be re-checked per site SOPs.
2. Received any investigational drug or used any investigational device within 30 days or 5 half-lives whichever is longer prior to the first dosing of study drug.
3. Clinically significant history of any serious drug sensitivity or allergy, or food allergy as determined by the Investigator (i.e., requiring epinephrine or steroids to treat).
4. Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders or abnormalities, or other major systemic disease that, according to the Investigator, would unduly risk the subject's safety or may impact the conduct of the study.
5. Presence of any disorder that would interfere with the swallowing, absorption, distribution, metabolism and excretion of the investigational product as judged by the Investigator. Surgery for appendicitis is acceptable.
6. Show evidence of significant active neuropsychiatric disease, including taking prescription medication for such diseases (including anti-depressant /anti-anxiety medication).
7. Presence of clinically significant physical, laboratory, or ECG findings at Screening that, in the opinion of the Investigator, may interfere with any aspect of study conduct or interpretation of results, or may present a safety issue to that particular subject. Laboratory results may be re-checked once per Investigator's discretion.
8. Liver function test results of aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≥ 1.25 upper limit of normal (ULN); with an exception of subjects considered eligible to participate in the study per Investigator's discretion.
9. History of vaso-vagal syncope within 5 years.
10. History of any major surgery within 6 months.
11. History of any active infection within 30 days prior to the first dosing.
12. Known history or positive test of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody (Ab), or human immunodeficiency virus type 1 (HIV-1) or 2 (HIV-2) Ab.
13. Subjects with a positive urine nicotine/cotinine test.
14. History of alcohol abuse as judged by the Investigator within approximately 1 year prior to admission. Average weekly alcohol intake > 14 units/week or are unwilling to stop alcohol consumption from 72 hr prior to dosing and outpatient visits and throughout the in-house periods until discharged from the clinical research unit and are unwilling to limit alcohol consumption during outpatient periods. Positive alcohol test at Screening or admission (One unit of alcohol equals about 12 ounces of beer, 5 ounces of wine or 1.5 ounces of spirits).
15. History of illicit drug abuse, within approximately 1 year prior to admission or evidence of current use as judged by the Investigator. Positive drug test, including marijuana, at Screening or admission.
16. Donation or loss of > 500 mL of blood within 56 days prior to admission.
17. Chronic use of prescription or non-prescription drugs (including vitamins and dietary or herbal supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) prior to the first dosing per Investigator's discretion.
18. Unable to comply with the safety monitoring requirements of this clinical study or is considered by the Investigator to be an unsuitable candidate for the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Up to Day 14
Incidence and severity of clinical findings on physical examination | Up to Day 8
Change from baseline in vital signs: Blood pressure (Systolic/Diastolic) | Up to Day 8
Change from baseline in vital signs: Body temperature | Up to Day 8
Change from baseline in vital signs: Respiratory rate | Up to Day 8
Change from baseline in vital signs: Heart rate | Up to Day 8
Incidence and severity of clinical laboratory abnormalities | Up to Day 8
  Hematology, serum chemistry and urinalysis
Change from baseline in 12-lead ECG parameters | Up to Day 8
  PR, QRS, QT and QTc intervals

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) for IA-14069 | Up to Day 8
Time to maximum concentration (Tmax) for IA-14069 | Up to Day 8
Area under the concentration-time curve (AUC) for IA-14069 | Up to Day 8
Terminal elimination half-life (t1/2) for IA-14069 | Up to Day 8
Apparent clearance (CL/F) for IA-14069 | Up to Day 8
Apparent volume of distribution (Vd/F) for IA-14069 | Up to Day 8
Pharmacokinetic (PK) in Food effect measured by Cmax for IA-14069 | Up to Day 8
PK in Food effect measured by Tmax for IA-14069 | Up to Day 8
PK in Food effect measured by AUC for IA-14069 | Up to Day 8
PK in Food effect measured by t1/2 for IA-14069 | Up to Day 8

OTHER OUTCOMES:
Change from baseline in concentration of Tumor necrosis factor in blood | Up to Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- ICON plc., Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No